CLINICAL TRIAL: NCT00465907
Title: Phase II Study of Weekly Paclitaxel, Carboplatin and Irinotecan in Patients With Advanced Non-Small Cell Lung Cancer Nad Malignant Pleural Effusion
Brief Title: Study of Weekly Paclitaxel, Carboplatin and Irinotecan to Treat Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS 0312; NA_00037282 (Other: JHM IRB)
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Lung Cancer
Keywords: lung cancer with malignant pleural effusion
MeSH Terms: conditions — Lung Neoplasms | interventions — Paclitaxel; Carboplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel, Carboplatin and Irinotecan (Experimental): Study of Weekly Paclitaxel, Carboplatin and Irinotecan in patients with Non-Small Cell Lung Carcinoma
  Interventions: Drug: Paclitaxel, Carboplatin and Irinotecan

INTERVENTIONS:
Drug: Paclitaxel, Carboplatin and Irinotecan — Paclitaxel-60mg/m2 weekly for 3 weeks Carboplatin - AUC 1.5, weekly for 3 weeks Irinotecan - 60mg/m2, weekly for 3 weeks

SUMMARY:
Evaluate the efficacy and toxicity of the weekly combination chemotherapy of Paclitaxel, Carboplatin and Irinotecan in Stage IIIb and IV NSCLC with malignant pleural effusion

DETAILED DESCRIPTION:
Lung cancer is the leading cancer death in many countries of the world including Singapore. Non-small cell lung cancer (NSCLC) consists of 80-85% of lung cancers, and is a major health problem. The main etiology of lung cancer is well recognized and established to be cigarette smoking which accounts for up to 80% of the cases in the western countries. Due to success of anti-smoking campaign, we anticipate to see less smoking related lung cancer and more non-smoking related lung cancer which is rising rapidly. For eg, currently in Singapore, smoking only accounts for 50-60% of all lung cancers, this is particularly true in female patients, as smoking occured in 30-40% of female lung cancer patients only.

It is unclear if there is any significant difference in the fundamental biology between smoking and non-smoking related lung cancers, particularly in areas of natural course of disease, genetic changes of tumor cells, clinical presentation, response to treatment or survival. These are potential aspects for further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of non-small cell lung cancer.
* Malignant pleural effusion proven by cytological examination.
* Patient must have stage IIIB or IV disease with malignant pleural effusion.
* We plan to recruit 16 patients who have smoked cigarettes of at least 20 pack per year, 16 patients who do not smoke but have been exposed to second hand smoking by living with a person who has smoked 20 pack per year cigarette in the same household and 16 patients who are non-smokers (never smoked) and no second hand smoking exposure in the same household. The accrual will be stopped once the number of patients is reached in each group.
* ECOG PS 0, 1 or 2.
* Measurable disease (in addition to malignant pleural effusion).
* No prior chemotherapy for metastatic or recurrent disease. Patient may have surgery or radiation or combined chemoradiation, or neoadjuvant chemotherapy at primary diagnosis. This kind of chemotherapy will not be counted as patient has had prior chemotherapy for metastatic or recurrent NSCLC.
* WBC > 3500/uL and ANC > 2,000/uL, platelet > 100,000/uL AST/ALT < 3 X UNL, bilirubin < 1.5 mg/dL ( or < 35 uM), creatinine < 1.5 mg/dL (or < 125uM for men and 90uM for women).
* Age > 18
* No history of congestive heart failure, myocardial infarction or life-threatening arrhythmia (such as ventricular tachycardia, supraventricular tachycardia, brachycardia < 40/min or atrial fibrillation or flutter with ventricular rate > 150/min) within 6 months of entry.
* Signed informed consent
* Negative mammogram and ovaries examination by CT scans and no history of breast cancer or ovarian cancer in female patients.
* Negative pregnancy test in female menstruating patient within one week of starting chemotherapy and use of effective contraceptive methods during study.
* Patients with brain metastasis will be eligible provided their neurological abnormality is stable or improved after whole brain radiation, stereostatic radiosurgery or gamma knife treatment and/or dexamethasone for 3 weeks and patients fulfil all other eligibility criteria.

Exclusion Criteria:

* ECOG performance status 3 or worse.
* Any prior chemotherapy regimen for metastatic or recurrent diseases.
* No measurable disease, even after drainage of pleural effusion.
* ANC < 1,999/uL or Bilirubin > 1.5 mg/dL (or > 35uM)
* Plt < 100,000/uL or
* ALT/AST > 3 x UNL
* Creatinine > 1.5mg/dL (or > 125uM)

Patient has history of congestive heart failure, myocardial infarction or life-threatening arrhythmia (such as ventricular tachycardia, supraventricular tachycardia, atrial fibrillation/flutter with ventricular rate > 150/min or bradycardia < 40/min) within 6 months before entry.

Prior history of breast cancer or ovarian cancer in female patients or any cancer except cured cervical carcinoma in-situ or skin cancer.

Fasting blood sugar > 200 mg/dL (> 14uM) except in patients on dexamethasone for brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-05; Primary Completion 2008-03 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and toxicity of the weekly combination chemotherapy of paclitaxel, carboplatin and irinotecan in Stage IIIB and IV NSCLC patients with malignant pleural effusion | 3 years

SECONDARY OUTCOMES:
To determine the pharmacokinetics and pharmacodynamics of paclitaxel and irinotecan in the blood and pleural effusion. | 3 years
To compare the gene expression pattern of non-small cell lung cancer from cigarette-smoking, passive smoking and no tobacco exposure patients before and after chemotherapy. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chang, MD, Principal Investigator — Johns Hopkins Singapore
Locations (1):
- Johns Hopkins Singapore International Medical Center, Singapore, Singapore